CLINICAL TRIAL: NCT04590963
Title: A Phase 3 Randomized, Double-blind, Multicenter, Global Study of Monalizumab or Placebo in Combination With Cetuximab in Participants With Recurrent or Metastatic Squamous Cell Carcinoma of the Head and Neck Previously Treated With an Immune Checkpoint Inhibitor
Brief Title: Assessment of Efficacy and Safety of Monalizumab Plus Cetuximab Compared to Placebo Plus Cetuximab in Recurrent or Metastatic Head and Neck Cancer
Acronym: INTERLINK-1
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Innate Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D7310C00001; 2024-511813-39-00 (Registry Identifier: CTIS (EU)); 2019-004770-25 (EudraCT Number)
Record Dates: First submitted 2020-09-23; First posted 2020-10-19 (Actual); Results first posted 2023-11-18 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-11

CONDITIONS: Squamous Cell Carcinoma of the Head and Neck
Keywords: head and neck cancer; Squamous Cell Carcinoma of the Head and Neck; monalizumab; cetuximab; Erbitux; oral cavity; larynx; pharynx; natural killer; oropharynx; hypopharynx
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Head and Neck Neoplasms; Laryngeal Diseases | interventions — monalizumab; Cetuximab

STUDY DESIGN:
Intervention Model Description: Parallel study. Participants will be randomized in a 2:1 ratio to monalizumab and cetuximab or placebo and cetuximab.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double blinded study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Monalizumab 750 mg Q2W + Cetuximab 400 mg/m^2 (Experimental): Participants will receive intravenous (IV) monalizumab 750 mg every two weeks (Q2W) and IV cetuximab 400 mg/m^2 initial dose followed by 250 mg/m^2 every one week (Q1W) until disease progression, unacceptable toxicity, withdrawal of consent, or another discontinuation criterion was met.
  Interventions: Drug: Monalizumab; Drug: Cetuximab
- Placebo Q2W + Cetuximab 400 mg/m^2 (Active Comparator): Participants will receieve IV placebo matched to monalizumab Q2W and IV cetuximab 400 mg/m^2 initial dose followed by 250 mg/m^2 Q1W until disease progression, unacceptable toxicity, withdrawal of consent, or another discontinuation criterion was met.
  Interventions: Drug: Cetuximab; Other: Placebo

INTERVENTIONS:
Drug: Monalizumab — Participants will receive IV infusion of monalizumab as stated in arm description.
  Other Names: IPH2201
  Arms: Monalizumab 750 mg Q2W + Cetuximab 400 mg/m^2
Drug: Cetuximab — Participants will receive IV infusion of cetuximab as stated in arm description.
  Other Names: Erbitux
Other: Placebo — Participants will receive IV infusion of placebo as stated in arm description.
  Arms: Placebo Q2W + Cetuximab 400 mg/m^2

SUMMARY:
This is a randomized, double-blind, multicenter, global Phase 3 study to assess the efficacy and safety of monalizumab and cetuximab, compared to placebo and cetuximab, in Participants with recurrent or metastatic head and neck cancer.

DETAILED DESCRIPTION:
Participants with recurrent or metastatic squamous cell carcinoma of the head and neck (SCCHN) who had prior immune checkpoint inhibitor and platinum-based chemotherapy treatment will be randomized in a 2:1 ratio to monalizumab and cetuximab or placebo and cetuximab. Efficacy and safety assessments will be performed periodically from the time of enrollment and throughout the study. Participants in all arms will continue therapy until progression, unacceptable toxicity, withdrawal of consent, or another discontinuation criterion is met. All Participants will be followed for survival after progression is confirmed.

ELIGIBILITY:
Inclusion Criteria:

* Are aged 18 years and over
* Recurrent or metastatic squamous cell carcinoma of the SCCHN, oral cavity, oropharynx, hypopharynx, or larynx which has progressed on or after previous systemic cancer therapy and is not amenable to curative therapy
* Received prior treatment using a programmed cell death ligand-1 (PD-L1) inhibitor
* Prior platinum failure
* Received 1 or 2 prior systemic regimens for recurrent or metastatic SCCHN
* Has measurable disease per RECIST 1.1
* A fresh or recently acquired tumor tissue for the purpose of biomarker testing
* World Health Organization (WHO)/ Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1

Exclusion Criteria:

* Head and neck cancer of any primary anatomic location in the head and neck not specified in the inclusion criteria, including participants with SCCHN of unknown primary or non-squamous histologies
* Had prior cetuximab therapy (unless it was administered in curative locally advanced setting with radiotherapy and no disease progression for at least 6 months following the last cetuximab dose)
* Active or prior documented autoimmune or inflammatory disorders (including inflammatory bowel disease [eg, colitis or Crohn's disease], diverticulitis
* Any concurrent anticancer treatment, except for hormonal therapy for non-cancer-related conditions (eg, hormone replacement therapy)

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 370 (Actual)
Dates: Start 2020-10-02 (Actual); Primary Completion 2022-05-11 (Actual); Study Completion 2026-09-24 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Roger B Cohen, MD, Principal Investigator — Abramson Cancer Center, Perelman Center for Advanced Medicine; Jérôme Fayette, MD, Principal Investigator — Centre Leon Berard; Dario Ruscica, MD, Study Director — AstraZeneca, Cambridge, UK
Locations (108):
- United States (16):
  - Research Site, Tucson, Arizona
  - Research Site, Chicago, Illinois
  - Research Site, Westwood, Kansas
  - Research Site, Boston, Massachusetts
  - Research Site, Ann Arbor, Michigan
  - Research Site, Rochester, Minnesota
  - Research Site, St Louis, Missouri
  - Research Site, Las Vegas, Nevada
  - Research Site, New York, New York
  - Research Site, Charlotte, North Carolina
  - Research Site, Winston-Salem, North Carolina
  - Research Site, Columbus, Ohio
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Pittsburgh, Pennsylvania
  - Research Site, Dallas, Texas
  - Research Site, Houston, Texas
- Research Site, CABA, Argentina
- Australia (4):
  - Research Site, Camperdown
  - Research Site, Elizabeth Vale
  - Research Site, Heidelberg
  - Research Site, Melbourne
- Research Site, Linz, Austria
- Belgium (4):
  - Research Site, Brussels
  - Research Site, Leuven
  - Research Site, Namur
  - Research Site, Roeselare
- Brazil (4):
  - Research Site, Belo Horizonte
  - Research Site, Porto Alegre
  - Research Site, Rio de Janeiro
  - Research Site, São Paulo
- Bulgaria (3):
  - Research Site, Panagyurishte
  - Research Site, Plovdiv
  - Research Site, Sofia
- Canada (4):
  - Research Site, Victoria, British Columbia
  - Research Site, Hamilton, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, Montreal, Quebec
- France (8):
  - Research Site, Avignon
  - Research Site, Bordeaux
  - Research Site, Clermont-Ferrand
  - Research Site, Dijon
  - Research Site, Lyon
  - Research Site, Marseille
  - Research Site, Montpellier
  - Research Site, Strasbourg
- Germany (7):
  - Research Site, Berlin
  - Research Site, Essen
  - Research Site, Freiburg im Breisgau
  - Research Site, Hanover
  - Research Site, Leipzig
  - Research Site, Ulm
  - Research Site, Würzburg
- Greece (3):
  - Research Site, Athens
  - Research Site, Chaïdári
  - Research Site, Thessaloniki
- Italy (7):
  - Research Site, Brescia
  - Research Site, Candiolo
  - Research Site, Florence
  - Research Site, Milan
  - Research Site, Modena
  - Research Site, Napoli
  - Research Site, Padua
- Japan (11):
  - Research Site, Chūōku
  - Research Site, Fukuoka
  - Research Site, Hiroshima
  - Research Site, Isehara-shi
  - Research Site, Kashiwa
  - Research Site, Kobe
  - Research Site, Kōtoku
  - Research Site, Okayama
  - Research Site, Sayama
  - Research Site, Sunto-gun
  - Research Site, Yokohama
- Netherlands (3):
  - Research Site, Amsterdam
  - Research Site, Maastricht
  - Research Site, Nijmegen
- Philippines (3):
  - Research Site, Manila
  - Research Site, Pasig
  - Research Site, Quezon City
- Poland (3):
  - Research Site, Bialystok
  - Research Site, Bydgoszcz
  - Research Site, Poznan
- Portugal (3):
  - Research Site, Coimbra
  - Research Site, Porto
  - Research Site, Vila Nova de Gaia
- Russia (4):
  - Research Site, Moscow
  - Research Site, Moscow Region
  - Research Site, Obninsk
  - Research Site, Saint Petersburg
- South Korea (5):
  - Research Site, Busan
  - Research Site, Cheongju-si
  - Research Site, Goyang-si
  - Research Site, Seongnam-si
  - Research Site, Seoul
- Spain (3):
  - Research Site, Barcelona
  - Research Site, Madrid
  - Research Site, Valencia
- Switzerland (3):
  - Research Site, Basel
  - Research Site, Bern
  - Research Site, Lausanne
- Taiwan (4):
  - Research Site, Changhua
  - Research Site, Taichung
  - Research Site, Tainan
  - Research Site, Taipei
- United Kingdom (4):
  - Research Site, London
  - Research Site, Manchester
  - Research Site, Newcastle upon Tyne
  - Research Site, Sutton

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of the timelines, please refer to the disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool. Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- [Derived] Nowojewski A, Wheal A, Dott W, Ruscica D, Ghiorghiu S, Valastro B. Implementation of the Study Participant Feedback Questionnaire to understand participant experience in a phase 3 oncology clinical trial. BMJ Open. 2025 Oct 28;15(10):e094596. doi: 10.1136/bmjopen-2024-094596. PMID 41151963
- See also: Redacted Statistical Analysis Plan — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D7310C00001&attachmentIdentifier=57ba61fb-176b-437b-b4a5-239f03702813&fileName=d7310c00001-statistical-analysis-plan-v4-marked-for-redaction_Redacted_(2).pdf&versionIdentifier=
- See also: Redacted Study Protocol — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D7310C00001&attachmentIdentifier=1f05756c-a18a-4c03-aa8d-bcf3521ecc44&fileName=d7310c00001-CSP_version_2_and_3_-_redacted.pdf&versionIdentifier=
- See also: Redacted CSR synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D7310C00001&attachmentIdentifier=eaf67e5d-9180-42b0-a9f7-dd302e97ce53&fileName=d7310c00001-abbreviated-study-synopsis-marked-for-redaction_Redacted_(1).pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at study sites located in Argentina, Australia, Austria, Belgium, Brazil, Bulgaria, Canada, France, Germany, Greece, Italy, Japan, Netherlands, Philippines, Poland, Portugal, Republic of Korea, Russia, Spain, Switzerland, Taiwan, United Kingdom, and United States of America.
Pre-assignment Details: A total of 370 participants were randomized (All randomized participants [ARP] set) in this study of which 368 participants received treatment. The analyses presented in this report are based on a clinical efficacy data cut-off (DCO) date of 11May2022, and clinical safety DCO date of 01Sep2022.
Groups:
- Monalizumab 750 mg Q2W + Cetuximab 400 mg/m^2: Participants received intravenous (IV) monalizumab 750 mg every two weeks (Q2W) and IV cetuximab 400 mg/m^2 initial dose followed by 250 mg/m^2 every 1 week (Q1W) until disease progression, unacceptable toxicity, withdrawal of consent, or another discontinuation criterion was met.
- Placebo Q2W + Cetuximab 400 mg/m^2: Participants receieved IV placebo matched to monalizumab Q2W and IV cetuximab 400 mg/m^2 initial dose followed by 250 mg/m^2 Q1W until disease progression, unacceptable toxicity, withdrawal of consent, or another discontinuation criterion was met.
Period: Overall Study
Arm/Group | Monalizumab 750 mg Q2W + Cetuximab 400 mg/m^2 | Placebo Q2W + Cetuximab 400 mg/m^2
Started | 247 | 123
Treated | 246 | 122
Completed | 0 | 0
Not Completed | 247 | 123
Not completed — Death | 118 | 59
Not completed — Lost to Follow-up | 1 | 1
Not completed — Progressive disease | 0 | 1
Not completed — Study terminated by sponsor | 103 | 50
Not completed — Withdrawal by Subject | 15 | 8
Not completed — Ongoing at data cut-off | 9 | 4
Not completed — Screen failure | 1 | 0

BASELINE CHARACTERISTICS:
Population: Baseline analysis population included all participants randomized up to the safety DCO date of 01Sep2022.
Groups:
- Monalizumab 750 mg Q2W + Cetuximab 400 mg/m^2: Participants received IV monalizumab 750 mg Q2W and IV cetuximab 400 mg/m^2 initial dose followed by 250 mg/m^2 Q1W until disease progression, unacceptable toxicity, withdrawal of consent, or another discontinuation criterion was met.
- Total: Total of all reporting groups
Arm/Group | Monalizumab 750 mg Q2W + Cetuximab 400 mg/m^2 | Placebo Q2W + Cetuximab 400 mg/m^2 | Total
Number analyzed (Participants) | 247 | 123 | 370
Age, Continuous [Mean (Standard Deviation); unit: Years] | 62.0 (10.4) | 61.4 (9.6) | 61.8 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42 | 29 | 71
  Male | 205 | 94 | 299
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 12 | 5 | 17
  Not Hispanic or Latino | 223 | 114 | 337
  Unknown or Not Reported | 12 | 4 | 16
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 66 | 30 | 96
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 0 | 3
  White | 169 | 89 | 258
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 9 | 4 | 13

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS) in Human Papillomavirus (HPV)-Unrelated Analysis Set
Description: The OS is defined as time from the date of randomization until death due to any cause regardless of whether the participant withdraws from randomized therapy or receives another anti-cancer therapy (i.e. date of death or censoring - date of randomization + 1). The OS was analyzed using Kaplan-Meier technique. Statistical analysis was performed using P-value from a stratified log-rank test and hazard ratio (HR) and confidence intervals (CIs) from a stratified Cox proportional hazards model. Analyses were stratified on World Health Organization/ Eastern Cooperative Oncology Group performance status (WHO/ECOG PS) (0 or 1) and number of prior lines of therapy in recurrent or metastatic (R/M) setting (1 or 2).
Time Frame: Baseline (-28 to -1) through 17.5 months (maximum observed duration)
Population: The HPV-unrelated analysis set included all participants who were randomized at least 2 months before the 11May2022 DCO (i.e. on or before 11Mar2022) and were either oropharyngeal cancer (OPC) HPV negative or non OPC regardless of the HPV status.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Monalizumab 750 mg Q2W + Cetuximab 400 mg/m^2 | Placebo Q2W + Cetuximab 400 mg/m^2
Number analyzed (Participants) | 145 | 71
Months | 8.8 [6.9 to 10.4] | 8.6 [6.0 to 14.5]
Statistical Analysis 1: Comparison: Monalizumab 750 mg Q2W + Cetuximab 400 mg/m^2 vs Placebo Q2W + Cetuximab 400 mg/m^2; Test type: Superiority; p = 0.989, Log Rank; P-value was calculated using stratified log-rank test, adjusted for WHO/ECOG PS (0/1) and number of prior lines of therapy in R/M setting; Hazard Ratio (HR) = 1.00, 95% CI 2-sided [0.660 to 1.537] — HR and CIs were calculated using a stratified Cox proportional hazards model, adjusted for WHO/ECOG PS, and number of lines of prior therapy in R/M setting

2. Secondary Outcome: Overall Survival in Full Analysis Set (FAS)
Description: The OS is defined as time from the date of randomization until death due to any cause regardless of whether the participant withdraws from randomized therapy or receives another anti-cancer therapy (i.e. date of death or censoring - date of randomization + 1). The OS was analyzed using Kaplan-Meier technique. Statistical analysis was performed using P-value from a stratified log-rank test and HR and CIs from a stratified Cox proportional hazards model. Analyses were stratified on HPV status (OPC HPV positive or HPV-unrelated), WHO/ECOG PS (0 or 1) and number of prior lines of therapy in R/M setting (1 or 2).
Time Frame: Baseline (-28 to -1) through 17.5 months (maximum observed duration)
Population: The FAS included all participants randomized at least 2 months before the DCO 11May2022 (i.e. on or before 11Mar2022).
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Monalizumab 750 mg Q2W + Cetuximab 400 mg/m^2 | Placebo Q2W + Cetuximab 400 mg/m^2
Number analyzed (Participants) | 175 | 89
Months | 8.8 [6.9 to 10.8] | 8.9 [6.0 to 15.1]
Statistical Analysis 1: Comparison: Monalizumab 750 mg Q2W + Cetuximab 400 mg/m^2 vs Placebo Q2W + Cetuximab 400 mg/m^2; Test type: Superiority; p = 0.891, Log Rank; P-value was calculated using stratified log-rank test, adjusted for HPV status, WHO/ECOG PS (0/1) and number of prior lines of therapy in R/M setting; Hazard Ratio (HR) = 1.03, 95% CI 2-sided [0.704 to 1.528] — HR and CIs were calculated using a stratified Cox proportional hazards model, adjusted for HPV status, WHO/ECOG PS, and number of lines of prior therapy in R/M setting

3. Secondary Outcome: Progression-Free Survival (PFS) Per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 by Investigator Assessment in HPV-unrelated Analysis Set
Description: PFS per RECIST 1.1 as assessed by the investigator is defined as time from randomization until date of RECIST 1.1-defined radiological progressive disease (PD) or death regardless of whether participant withdraws from therapy or received subsequent anticancer therapy prior to progression. PD: at least 20% increase in sum of diameters of target lesions (TLs), taking as reference the smallest sum on study (nadir) and sum must demonstrate an absolute increase of at least 5 mm from nadir or unequivocal progression of existing non-TLs (NTLs) or appearance of new lesions. PFS was analyzed using Kaplan-Meier technique. Statistical analysis was performed using P-value from stratified log-rank test and HR and CIs from a stratified Cox proportional hazards model. Analyses were stratified on WHO/ECOG PS (0/1) and no. of prior lines of therapy in R/M setting.
Time Frame: Baseline (-28 to -1) through 17.5 months (maximum observed duration)
Population: The HPV-unrelated analysis set included all participants who were randomized at least 2 months before the 11May2022 DCO (i.e. on or before 11Mar2022) and were either OPC HPV negative or non OPC regardless of the HPV status.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Monalizumab 750 mg Q2W + Cetuximab 400 mg/m^2 | Placebo Q2W + Cetuximab 400 mg/m^2
Number analyzed (Participants) | 145 | 71
Months | 3.6 [3.1 to 3.7] | 3.8 [2.4 to 4.9]
Statistical Analysis 1: Comparison: Monalizumab 750 mg Q2W + Cetuximab 400 mg/m^2 vs Placebo Q2W + Cetuximab 400 mg/m^2; Test type: Superiority; p = 0.574, Log Rank; [statistical method as in outcome 1, analysis 1]; Hazard Ratio (HR) = 1.11, 95% CI 2-sided [0.790 to 1.568] — [estimate comment as in outcome 1, analysis 1]

4. Secondary Outcome: Progression-Free Survival Per RECIST 1.1 by Investigator Assessment in FAS
Description: PFS per RECIST 1.1 as assessed by the investigator is defined as time from randomization until date of RECIST 1.1-defined radiological progressive disease (PD) or death regardless of whether participant withdraws from therapy or received subsequent anticancer therapy prior to progression. PD: at least 20% increase in sum of diameters of target lesions (TLs), taking as reference the smallest sum on study (nadir) and sum must demonstrate an absolute increase of at least 5 mm from nadir or unequivocal progression of existing NTLs or appearance of new lesions. PFS was analyzed using Kaplan-Meier technique. Statistical analysis was performed using P-value from a stratified log-rank test and HR and CIs from a stratified Cox proportional hazards model. Analyses were stratified on HPV status, WHO/ECOG PS (0/1) and no. of prior lines of therapy in R/M setting.
Time Frame: Baseline (-28 to -1) through 17.5 months (maximum observed duration)
Population: The FAS included all participants randomized at least 2 months before the DCO 11May2022 (i.e. on or before 11Mar2022).
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Monalizumab 750 mg Q2W + Cetuximab 400 mg/m^2 | Placebo Q2W + Cetuximab 400 mg/m^2
Number analyzed (Participants) | 175 | 89
Months | 3.5 [2.3 to 3.7] | 3.7 [2.2 to 4.2]
Statistical Analysis 1: Comparison: Monalizumab 750 mg Q2W + Cetuximab 400 mg/m^2 vs Placebo Q2W + Cetuximab 400 mg/m^2; Test type: Superiority; p = 0.530, Log Rank; [statistical method as in outcome 2, analysis 1]; Hazard Ratio (HR) = 1.11, 95% CI 2-sided [0.818 to 1.512] — [estimate comment as in outcome 2, analysis 1]

5. Secondary Outcome: Percentage of Participants With Objective Response (OR) Per RECIST 1.1 in HPV-unrelated Analysis Set
Description: The OR is defined as the percentage of participants with at least one confirmed investigator-assessed response of complete response (CR) or partial response (PR) as assessed by RECIST 1.1 guidelines. The CR is defined as disappearance of all TLs and NTLs, any pathological lymph nodes (target and non-target) must have reduction in short axis < 10 mm, and no new lesions. The PR is defined as at least a 30% decrease in the sum of the diameters (SoD) of TLs (compared to baseline) and no new lesions. Confirmation of CR and PR is required by a repeat, consecutive assessment no less than 4 weeks from the date of first documentation. Percentage of participants with OR is reported. Participants who had measurable disease at baseline per the site investigator were analyzed for this outcome.
Time Frame: Baseline (-28 to -1) through 17.5 months (maximum observed duration)
Population: The HPV-unrelated analysis set included all participants who were randomized at least 2 months before the 11May2022 DCO (i.e. on or before 11Mar2022) and were either OPC HPV negative or non OPC regardless of the HPV status. Participants who had measurable disease at baseline per the site investigator were analyzed for this outcome.
Measure: Number; unit: Percentage of Participants
Arm/Group | Monalizumab 750 mg Q2W + Cetuximab 400 mg/m^2 | Placebo Q2W + Cetuximab 400 mg/m^2
Number analyzed (Participants) | 145 | 71
Percentage of Participants | 15.2 [0.274 to 1.154] | 23.9
Statistical Analysis 1: Comparison: Monalizumab 750 mg Q2W + Cetuximab 400 mg/m^2 vs Placebo Q2W + Cetuximab 400 mg/m^2; Test type: Superiority; p = 0.115, Regression, Logistic; P-value is based on twice the change in log-likelihood resulting from the addition of a treatment factor to the model; Odds Ratio (OR) = 0.56, 95% CI 2-sided [0.274 to 1.154] — The analysis was performed using a logistic regression model, with treatment as a covariate and adjusting for WHO/ECOG PS, and number of lines of prior therapy in the R/M setting with 95% CI calculated by profile likelihood

6. Secondary Outcome: Percentage of Participants With OR Per RECIST 1.1 in FAS
Description: The OR is defined as the percentage of participants with at least one confirmed investigator-assessed response of CR or PR as assessed by RECIST 1.1 guidelines. The CR is defined as disappearance of all TLs and NTLs, any pathological lymph nodes (target and non-target) must have reduction in short axis < 10 mm, and no new lesions. The PR is defined as at least a 30% decrease in the SoD of TLs (compared to baseline) and no new lesions. Confirmation of CR and PR is required by a repeat, consecutive assessment no less than 4 weeks from the date of first documentation. Percentage of participants with OR is reported. Participants who had measurable disease at baseline per the site investigator were analyzed for this outcome.
Time Frame: Baseline (-28 to -1) through 17.5 months (maximum observed duration)
Population: The FAS included all participants randomized at least 2 months before the DCO 11May2022 (i.e. on or before 11Mar2022). Participants who had measurable disease at baseline per the site investigator were analyzed for this outcome.
Measure: Number; unit: Percentage of Participants
Arm/Group | Monalizumab 750 mg Q2W + Cetuximab 400 mg/m^2 | Placebo Q2W + Cetuximab 400 mg/m^2
Number analyzed (Participants) | 175 | 89
Percentage of Participants | 13.1 [0.297 to 1.231] | 19.1
Statistical Analysis 1: Comparison: Monalizumab 750 mg Q2W + Cetuximab 400 mg/m^2 vs Placebo Q2W + Cetuximab 400 mg/m^2; Test type: Superiority; p = 0.162, Regression, Logistic; P-value is based on twice the change in log-likelihood resulting from the addition of a treatment factor to the model; Odds Ratio (OR) = 0.60, 95% CI 2-sided [0.297 to 1.231] — The analysis was performed using a logistic regression model, with treatment as a covariate and adjusting for HPV Status, WHO/ECOG PS, and number of lines of prior therapy in the R/M setting with 95% CI calculated by profile likelihood

7. Secondary Outcome: Duration of Response (DoR) Per RECIST 1.1 in HPV-unrelated Analysis Set
Description: The DoR is defined as the time from the date of first documented confirmed response until date of documented progression or death in the absence of disease progression (i.e. date of PFS event or censoring - date of first response + 1). The CR is defined as disappearance of all target and non-target lesions, no new lesions, and normalization of tumor marker level. The PR is defined as at least a 30% decrease in the SoDs of TLs (compared to baseline) and no new lesions. Confirmation of CR and PR is required by a repeat, consecutive assessment no less than 4 weeks from the date of first documentation. The PD is defined as at least a 20% increase in the SoDs of TLs, taking as reference the smallest previous SoDs (nadir) and the sum must demonstrate an absolute increase of at least 5 mm from nadir or unequivocal progression of existing NTLs or appearance of new lesions. The DoR was analyzed using Kaplan-Meier technique.
Time Frame: Baseline (-28 to -1) through 17.5 months (maximum observed duration)
Population: The HPV-unrelated analysis set included all participants who were randomized at least 2 months before the 11May2022 DCO (i.e. on or before 11Mar2022) and were either OPC HPV negative or non OPC regardless of the HPV status. The DoR is assessed for only those participants who had OR.
Measure: Median (Inter-Quartile Range); unit: Months
Arm/Group | Monalizumab 750 mg Q2W + Cetuximab 400 mg/m^2 | Placebo Q2W + Cetuximab 400 mg/m^2
Number analyzed (Participants) | 22 | 17
Months | 5.7 [5.5 to 8.1] | 5.6 [4.4 to NA] — The upper limit of 75th percentile was not reached because there were not enough responders who subsequently progressed or died in this treatment group.

8. Secondary Outcome: Duration of Response Per RECIST 1.1 in FAS
Description: as for outcome 7
Time Frame: Baseline (-28 to -1) through 17.5 months (maximum observed duration)
Population: The FAS included all participants randomized at least 2 months before the DCO 11May2022 (i.e. on or before 11Mar2022). The DoR is assessed for only those participants who had OR.
Measure: Median (Inter-Quartile Range); unit: Months
Arm/Group | Monalizumab 750 mg Q2W + Cetuximab 400 mg/m^2 | Placebo Q2W + Cetuximab 400 mg/m^2
Number analyzed (Participants) | 23 | 17
Months | 5.7 [5.3 to 8.1] | 5.6 [4.4 to NA] — The upper limit of 75th percentile was not reached because there were not enough responders who subsequently progressed or died in this treatment group.

9. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs)
Description: An adverse event (AE) is any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. TEAEs included events from the first dose of study drug, up to 90 days after the last dose of study drug received or up to the start date of any subsequent anticancer therapy following discontinuation of study drug, or the final safety DCO date of 01Sep2022, whichever occurred first.
Time Frame: Day 1 through 21.4 months (maximum observed duration)
Population: The Safety Analysis Set included all participants randomized at least 2 months before the DCO 01Sep2022 (i.e. on or before 01Jul2022).
Measure: Count of Participants; unit: Participants
Arm/Group | Monalizumab 750 mg Q2W + Cetuximab 400 mg/m^2 | Placebo Q2W + Cetuximab 400 mg/m^2
Number analyzed (Participants) | 246 | 122
Participants | 236 | 120

10. Secondary Outcome: Number of Participants With Abnormal Clinical Laboratory Parameters Reported as TEAEs
Description: Participants with abnormal laboratory parameters reported as TEAEs are reported. Laboratory analysis included hematology and clinical chemistry. TEAEs included events from the first dose of study drug, up to 90 days after the last dose of study drug received or up to the start date of any subsequent anticancer therapy following discontinuation of study drug, or the final safety DCO date of 01Sep2022, whichever occurred first.
Time Frame: Day 1 through 21.4 months (maximum observed duration)
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | Monalizumab 750 mg Q2W + Cetuximab 400 mg/m^2 | Placebo Q2W + Cetuximab 400 mg/m^2
Number analyzed (Participants) | 246 | 122
Participants
  Anaemia | 35 | 15
  Anaemia folate deficiency | 1 | 0
  Hypochromic anaemia | 1 | 0
  Iron deficiency anaemia | 1 | 0
  Leukocytosis | 3 | 2
  Leukopenia | 0 | 1
  Lymphocytosis | 0 | 1
  Lymphopenia | 3 | 1
  Neutropenia | 1 | 1
  Neutrophilia | 0 | 2
  Normocytic anaemia | 1 | 0
  Thrombocytopenia | 1 | 0
  Thrombocytosis | 1 | 2
  Hyperthyroidism | 0 | 1
  Hypoparathyroidism | 1 | 0
  Hypothyroidism | 15 | 7
  Hyperamylasaemia | 1 | 0
  Hypercalcaemia | 7 | 4
  Hyperglycaemia | 7 | 5
  Hyperkalaemia | 3 | 1
  Hyperlipasaemia | 1 | 0
  Hypermagnesaemia | 3 | 1
  Hyperphosphataemia | 1 | 0
  Hypoalbuminaemia | 2 | 4
  Hypocalcaemia | 11 | 4
  Hypoglycaemia | 1 | 0
  Hypokalaemia | 13 | 9
  Hypomagnesaemia | 42 | 21
  Hyponatraemia | 6 | 3
  Hypophosphataemia | 9 | 8
  Iron deficiency | 1 | 0
  Activated partial thromboplastin time prolonged | 1 | 0
  Alanine aminotransferase increased | 7 | 5
  Amylase increased | 6 | 3
  Aspartate aminotransferase increased | 7 | 4
  Blood alkaline phosphatase increased | 7 | 3
  Blood beta-D-glucan increased | 0 | 1
  Blood bilirubin increased | 3 | 0
  Blood creatine phosphokinase increased | 2 | 0
  Blood creatinine increased | 6 | 3
  Blood iron decreased | 0 | 1
  Blood lactate dehydrogenase increased | 3 | 3
  Blood phosphorus decreased | 1 | 0
  Blood potassium decreased | 1 | 0
  Blood thyroid stimulating hormone abnormal | 1 | 0
  Blood thyroid stimulating hormone increased | 2 | 3
  Blood urea increased | 0 | 1
  C-reactive protein increased | 0 | 2
  Gamma-glutamyltransferase increased | 5 | 1
  Inflammatory marker increased | 1 | 0
  International normalised ratio increased | 1 | 0
  Lipase increased | 12 | 2
  Lymphocyte count decreased | 3 | 0
  Neutrophil count decreased | 2 | 3
  Neutrophil count increased | 1 | 0
  Platelet count decreased | 1 | 0
  Platelet count increased | 1 | 0
  Transaminases increased | 1 | 0
  White blood cell count decreased | 2 | 3
  White blood cell count increased | 1 | 0
  Dyslipidaemia | 0 | 1

11. Secondary Outcome: Number of Participants With Abnormal Vital Signs Reported as TEAEs
Description: Participants with abnormal vital signs (heart rate, blood pressure, temperature, and respiratory rate) reported as TEAEs are reported. TEAEs included events from the first dose of study drug, up to 90 days after the last dose of study drug received or up to the start date of any subsequent anticancer therapy following discontinuation of study drug, or the final safety DCO date of 01Sep2022, whichever occurred first.
Time Frame: Day 1 through 21.4 months (maximum observed duration)
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | Monalizumab 750 mg Q2W + Cetuximab 400 mg/m^2 | Placebo Q2W + Cetuximab 400 mg/m^2
Number analyzed (Participants) | 246 | 122
Participants
  Hypertension | 4 | 4
  Hypotension | 11 | 3
  Hypoxia | 0 | 1
  Hyperpyrexia | 1 | 0
  Pyrexia | 18 | 10

12. Secondary Outcome: Number of Participants With Electrocardiograms (ECGs) Reported as TEAEs
Description: Participants with Abnormal ECGs reported as TEAEs are reported. TEAEs included events from the first dose of study drug, up to 90 days after the last dose of study drug received or up to the start date of any subsequent anticancer therapy following discontinuation of study drug, or the final safety DCO date of 01Sep2022, whichever occurred first.
Time Frame: Day 1 through 21.4 months (maximum observed duration)
Population: The Safety Analysis Set (SAS) included all participants randomized at least 2 months before the DCO 01Sep2022 (i.e. on or before 01Jul2022).
Measure: Count of Participants; unit: Participants
Arm/Group | Monalizumab 750 mg Q2W + Cetuximab 400 mg/m^2 | Placebo Q2W + Cetuximab 400 mg/m^2
Number analyzed (Participants) | 246 | 122
Participants
  Electrocardiogram QT prolonged | 1 | 0
  Arrhythmia | 0 | 1
  Atrial fibrillation | 1 | 0
  Sinus tachycardia | 2 | 0
  Tachycardia | 2 | 2
  Ventricular arrhythmia | 0 | 1

ADVERSE EVENTS:
Time Frame: Day 1 through 21.4 months (maximum observed duration)
Description: All-Cause Mortality (ACM) reports data for ARP set; AE/SAE data is reported for SAS. Two participants died in follow-up period in each arm, after consent withdrawal from study, so number of deaths reported in ACM is different than of participant flow. TEAEs: Events from first dose of study drug (SD) up to 90 days after last dose of SD received or up to start date of any subsequent anticancer therapy following discontinuation of SD or final safety DCO of 01Sep22, whichever occurred first.
Arm/Group | Monalizumab 750 mg Q2W + Cetuximab 400 mg/m^2 | Placebo Q2W + Cetuximab 400 mg/m^2
All-Cause Mortality (participants affected / at risk) | 120/247 | 61/123
Serious Adverse Events (participants affected / at risk) | 77/246 | 27/122
Other Adverse Events (participants affected / at risk) | 213/246 | 111/122
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Monalizumab 750 mg Q2W + Cetuximab 400 mg/m^2 (N=246) | Placebo Q2W + Cetuximab 400 mg/m^2 (N=122)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Stevens-johnson syndrome (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
Venous thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Duodenal ulcer (Gastrointestinal disorders) | 1 (1) | 1 (1)
Faecaloma (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haematemesis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal ischaemia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Mouth haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 3 (3) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Death (General disorders) | 1 (1) | 1 (1)
General physical health deterioration (General disorders) | 1 (1) | 0 (0)
Malaise (General disorders) | 1 (1) | 0 (0)
Mucosal inflammation (General disorders) | 1 (1) | 0 (0)
Pain (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 4 (4) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 2 (2) | 0 (0)
Cytokine release syndrome (Immune system disorders) | 1 (1) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 1 (1)
Hypersensitivity (Immune system disorders) | 1 (1) | 0 (0)
Infusion related hypersensitivity reaction (Immune system disorders) | 2 (2) | 1 (1)
Arthritis bacterial (Infections and infestations) | 1 (1) | 0 (0)
Bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Covid-19 (Infections and infestations) | 5 (5) | 1 (1)
Covid-19 pneumonia (Infections and infestations) | 1 (1) | 1 (1)
Fungaemia (Infections and infestations) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 1 (1)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0)
Labyrinthitis (Infections and infestations) | 1 (1) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1)
Lung abscess (Infections and infestations) | 1 (1) | 0 (0)
Osteomyelitis (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 13 (15) | 8 (9)
Pneumonia aspiration (Infections and infestations) | 3 (3) | 1 (1)
Pneumonia pseudomonal (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 4 (5) | 0 (0)
Septic shock (Infections and infestations) | 0 (0) | 1 (1)
Cardiac tamponade (Cardiac disorders) | 1 (1) | 0 (0)
Staphylococcal infection (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 2 (2) | 3 (3)
Post procedural complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Lipase increased (Investigations) | 1 (1) | 0 (0)
Urine output decreased (Investigations) | 1 (1) | 0 (0)
White blood cell count decreased (Investigations) | 1 (1) | 0 (0)
Acidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypophagia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Blindness unilateral (Eye disorders) | 0 (0) | 1 (1)
Sacral pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Pachymeningitis (Nervous system disorders) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 1 (1) | 1 (1)
Syncope (Nervous system disorders) | 2 (2) | 0 (0)
Colitis ulcerative (Gastrointestinal disorders) | 1 (1) | 0 (0)
Mental status changes (Psychiatric disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 1 (1)
Chronic kidney disease (Renal and urinary disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Laryngeal haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Pharyngeal haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pharyngeal swelling (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (3) | 2 (2)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Thoracic haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Tracheal inflammation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Monalizumab 750 mg Q2W + Cetuximab 400 mg/m^2 (N=246) | Placebo Q2W + Cetuximab 400 mg/m^2 (N=122)
Diarrhoea (Gastrointestinal disorders) | 27 (32) | 14 (17)
Pruritus (Skin and subcutaneous tissue disorders) | 32 (35) | 18 (21)
Rash (Skin and subcutaneous tissue disorders) | 56 (60) | 27 (29)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 9 (9) | 7 (8)
Skin fissures (Skin and subcutaneous tissue disorders) | 16 (21) | 9 (9)
Nausea (Gastrointestinal disorders) | 26 (32) | 20 (24)
Stomatitis (Gastrointestinal disorders) | 31 (33) | 16 (18)
Vomiting (Gastrointestinal disorders) | 23 (27) | 9 (12)
Anaemia (Blood and lymphatic system disorders) | 33 (42) | 15 (17)
Asthenia (General disorders) | 19 (19) | 9 (12)
Fatigue (General disorders) | 48 (53) | 20 (24)
Pyrexia (General disorders) | 15 (17) | 10 (10)
Covid-19 (Infections and infestations) | 7 (7) | 7 (7)
Conjunctivitis (Infections and infestations) | 7 (8) | 7 (7)
Paronychia (Infections and infestations) | 28 (29) | 19 (22)
Infusion related reaction (Injury, poisoning and procedural complications) | 21 (23) | 12 (14)
Weight decreased (Investigations) | 14 (16) | 6 (7)
Hypothyroidism (Endocrine disorders) | 15 (17) | 7 (8)
Decreased appetite (Metabolism and nutrition disorders) | 16 (16) | 15 (15)
Hypokalaemia (Metabolism and nutrition disorders) | 13 (18) | 9 (12)
Hypomagnesaemia (Metabolism and nutrition disorders) | 42 (47) | 20 (29)
Hypophosphataemia (Metabolism and nutrition disorders) | 9 (10) | 8 (8)
Dizziness (Nervous system disorders) | 15 (16) | 5 (5)
Headache (Nervous system disorders) | 18 (19) | 7 (9)
Cough (Respiratory, thoracic and mediastinal disorders) | 17 (18) | 6 (6)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 17 (20) | 5 (5)
Constipation (Gastrointestinal disorders) | 33 (36) | 11 (11)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 80 (90) | 42 (49)
Dry skin (Skin and subcutaneous tissue disorders) | 28 (28) | 14 (16)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 13 (13) | 7 (9)

LIMITATIONS AND CAVEATS:
Study enrolment was discontinued after the planned initial interim futility analysis (IA1) due to unlikelihood of achieving statistical significance for OS in the primary endpoint (HPV-unrelated). Therefore, symptoms, function, health-related quality of life (HRQoL), European Organization for Research and Treatment of Cancer (EORTC) scale/item score, pharmacokinetic (PK) parameters, immunogenicity, human leukocyte antigen E (HLA-E), and NKp46+ expression outcomes were not evaluated.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
MedImmune has 60 days to review results communications prior to public release and may delete information that compromises ongoing studies or is considered proprietary. This restriction is not intended to compromise the objective scientific integrity of the manuscript, it being understood that results shall be published regardless of outcome.

DOCUMENTS (2):
  • Study Protocol (2021-07-07): https://cdn.clinicaltrials.gov/large-docs/63/NCT04590963/Prot_000.pdf
  • Statistical Analysis Plan (2022-07-19): https://cdn.clinicaltrials.gov/large-docs/63/NCT04590963/SAP_001.pdf